CLINICAL TRIAL: NCT07169552
Title: A Multicenter, Single-arm, Open-label Phase II Clinical Study to Evaluate the Efficacy and Safety of HC010 for Injection in the First-line Treatment of Advanced Non-small Cell Lung Cancer Positive for Programmed Death Ligand-1 (PD-L1)
Brief Title: HC010 in First-line PD-L1 Positive Advanced NSCLC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HC Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-HC010-201
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HC010 (Experimental)
  Interventions: Drug: HC010

INTERVENTIONS:
Drug: HC010 — HC010 Q3W intravenous infusion

SUMMARY:
Phase 2 clinical study to evaluate the efficacy, safety, pharmacokinetics and immunogenicity profile of HC010 for injection in patients with positive PD-L1 (TPS ≥1%)

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label Phase 2 clinical study to evaluate the efficacy, safety, pharmacokinetics and immunogenicity profile of HC010 for injection as monotherapy in first-line treatment of locally advanced or metastatic non-small cell lung cancer with positive PD-L1 (TPS ≥1%), negative EGFR mutations and negative ALK.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in the study, communicate well with investigators, understand and voluntarily complete the study process according to this protocol, and sign the informed consent form (ICF).
* 2. Male or female, aged ≥ 18 years at the time of signing the informed consent form.
* 3. Histologically or cytologically confirmed locally advanced or metastatic (stage IIIb~IV) NSCLC (United States Cancer Confederation [AJCC] 8th edition), positive PD-L1 expression confirmed by IHC with central laboratory or local test results.
* 4. Not previously receiving systemic therapy for locally advanced or metastatic NSCLC; not allowed if the last dose of prior treatment is <6 months from disease recurrence in subjects who received prior adjuvant or neoadjuvant therapy.
* 5. No EGFR mutation/ROS1 rearrangement/ALK rearrangement. If other targeted mutations such as BRAF V600E mutation/NTRK1/2/3 gene fusion/MET14 exon skipping mutation/RET rearrangement positive are known, they will not be included in this study if the corresponding targeted therapy drugs have been approved.
* 6. Expected survival ≥ 3 months.
* 7.There should be at least one measurable lesion according to RECIST v1.1; radiotherapy-experienced lesions may not be selected as target lesions, unless the radiotherapy lesion is the only measurable lesion and clearly progresses based on imaging judgment.
* 8. Eastern Cooperative Oncology Group (ECOG) performance status scored 0 or 1 in the United States and did not worsen within one week prior to first dose.
* 9. Subjects (both female and male) agreed to use effective contraception from signing the ICF until 180 days after last dose of investigational product. Female patients of childbearing potential must have a negative blood or urine pregnancy test within 7 days prior to the first dose; females who are not pregnant or lactating from signing informed consent until 6 months after the last use of investigational drug (including those who agree to stop breastfeeding during this period).

Exclusion Criteria:

* 1. Subjects who have received Chinese patent medicine or immunomodulatory drugs (including but not limited to thymopeptide, interferon and interleukin) with anti-tumor indications within 2 weeks before the first dose;
* 2. Pulmonary radiation therapy >30 Gy within 6 months prior to the first dose;
* 3. Complete palliative radiotherapy within 7 days before the first dose;
* 4. Any other form of anti-tumor therapy is expected to be required during the study;
* 5. Pericardial effusion (a stable small amount of pericardium can be included actively), or uncontrolled or symptomatic pleural and ascites effusions requiring puncture drainage;
* 6. Presence of brain stem, meningeal metastases/meningitis carcinoma, spinal cord metastasis or compression;
* 7. Known brain metastases. Previously treated subjects with brain metastasis may participate in the study if they are clinically stable for at least 4 weeks prior to first dose, have no evidence of new or expanded brain metastases, and discontinue steroids 7 days prior to first dose. According to this definition, the stability of brain metastasis should be established prior to the first dose of study drug. Subjects with known untreated asymptomatic brain metastases stable for at least 4 weeks (i.e., no neurological symptoms, no corticosteroid treatment required, no or only slight peripheral edema, no lesion >1.5 cm, or stable brain lesion as determined by imaging) can participate in the study;
* 8. Patients who have taken systemic corticosteroids (> 10 mg prednisone or equivalent daily) or other immunosuppressive drugs (such as cyclophosphamide, azathioprine, methotrexate, thalidomide, TNF-α inhibitors, etc.) within 2 weeks prior to the first dose;
* 9. Systemic infection or other serious infection requiring intravenous antibiotics for >7 days within 2 weeks prior to the first dose, or fever of unexplained origin >38.5 °C during screening and before enrollment (except for fever due to tumor in the investigator's judgment).
* 10. Concurrent with other malignant tumors within 5 years before the first dose, except for patients with adequately treated cervical carcinoma in situ, basal cell, squamous epithelial cell skin cancer, papillary thyroid carcinoma, local prostate cancer after radical resection and ductal carcinoma in situ after radical resection;
* 11. Subjects with diseases that may jeopardize their safety or compliance with the study protocol, and other conditions unsuitable for participation in this study as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 24months
  Objective response rate (ORR) assessed by the investigator according to RECIST 1.1 criteria;

SECONDARY OUTCOMES:
Safety and tolerability | 24 months
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.
DCR | 24 months
  Disease control rate (DCR), which is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
DoR | 24 months
  Duration of response (DoR), which is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
PFS | 24 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first assessed by investigator Per RECIST 1.1.
OS | 24 months
  Overall Survival (OS) in the ITT population

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No